CLINICAL TRIAL: NCT02668432
Title: Use of Amiodarone in Atrial Fibrillation Associated With Severe Sepsis or Septic Shock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20150864H
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-11

CONDITIONS: New Onset Atrial Fibrillation; Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Partial Load (Experimental): All patients will receive a 150 mg intravenous (IV) bolus dose of amiodarone, followed immediately by a continuous infusion of 1 mg/min for the first six hours, with a recommended reduction to 0.5 mg/min subsequently. Conversion from IV to oral (PO) amiodarone will occur based on patient hemodynamic stability and physician/pharmacist discretion. Patients randomized to the partial load arm will receive <4g IV or < 8g PO. The assigned total loading dose will include all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO amount (accounting for 50% bioavailability of PO versus IV amiodarone).
  Interventions: Drug: Amiodarone
- Full Load (Active Comparator): All patients will receive a 150 mg intravenous (IV) bolus dose of amiodarone, followed immediately by a continuous infusion of 1 mg/min for the first six hours, with a recommended reduction to 0.5 mg/min subsequently. Conversion from IV to oral (PO) amiodarone will occur based on patient hemodynamic stability and physician/pharmacist discretion. Patients randomized to the partial load arm will receive (≥ 5g IV or ≥10g PO +/- 20%). The assigned total loading dose will include all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO amount (accounting for 50% bioavailability of PO versus IV amiodarone).
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — Patients will receive a 150 mg IV bolus amiodarone dose, followed by a 1 mg/min continuous infusion for six hours, then 0.5 mg/min. Conversion to PO amiodarone will be based on patient hemodynamic stability and physician/pharmacist discretion. The total loading dose will be calculated based on all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO equivalents (accounting for 50% bioavailability of PO vs IV amiodarone). Randomization may be overridden by the attending or fellow physician if the patient's severity of illness warrants. Discontinuation of amiodarone in the full-load group will be at the discretion of the physician/pharmacists, after the pre-determined randomization loading dose has been provided.
  Other Names: Cordarone; Pacerone

SUMMARY:
Purpose/Objectives: Severe sepsis and septic shock are a common cause of new onset atrial fibrillation (NOAF) in the intensive care unit. Development of NOAF in this setting can prolong length of stay and increase mortality. Amiodarone is the most commonly used agent used in this setting to control rate and rhythm. However, limited data exist detailing appropriate dosing in this setting. The primary objective of this study is to evaluate two amiodarone dosing strategies, a full loading dose versus a partial loading dose, in patients with new-onset atrial fibrillation (AF) due to severe sepsis or septic shock to assess the mean heart rate every 6 hours after initiation of amiodarone infusion to day 7 or death.

Research Design/Plan: Consecutive patients admitted to the medical or cardiac intensive care unit at University Hospital with NOAF in the setting of severe sepsis or septic shock will be screened for study inclusion. Data will be collected and stored using Microsoft Excel or Access and analyzed with JMP 12.0 and SPSS.

Methods: Patients aged 18 years or older who develop new-onset atrial fibrillation in the setting of severe sepsis or septic shock and in whom the medical team deems appropriate to initiate amiodarone therapy in will be considered for study inclusion. Patients will receive intravenous (IV) and oral (PO) amiodarone, as per the standard of care. Patients will be randomized to a certain quantitative loading dose strategy; either a full loading dose (≥ 5g IV or ≥10g PO +/- 20%) or a partial loading dose (<4g IV or < 8g PO).

Clinical Relevance: With intensive care unit length of stay (ICU LOS) and mortality being twice as high in NOAF with sepsis as compared to septic patients without NOAF, the investigators ultimately aim to identify a management strategy that may minimize this morbidity and mortality while also minimizing exposure to a drug that may cause serious adverse effects.

DETAILED DESCRIPTION:
Step-by-Step Methods:

Population: The study will be conducted at University Hospital, the 716-bed county hospital for Bexar County and serves a varied population, including patients from medically underserved areas. The patient population will come from the medical intensive care unit and the cardiac intensive care unit, a 20 and 26-bed unit, respectively, at University Hospital that is the clinical practice and teaching site for one study investigator.

Screening: Consecutive patients admitted to the medical or cardiac intensive care unit at University Hospital with new onset atrial fibrillation in the setting of severe sepsis or septic shock will be screened for study inclusion. Participants will be 18 years or older. Patients who develop new-onset atrial fibrillation in the setting of severe sepsis or septic shock will be considered for study inclusion. Exclusion criteria apply to those younger than 18 years of age, those with a history of atrial flutter, baseline QTc (a measurement made on a electrocardiogram which measures the start of the Q wave to the end of the T wave) > 500 msec, atrial fibrillation during the index admission or in their past medical history, second or third degree atrioventricular (AV) block, those recovering from cardiac surgery done during the same hospital admission, those who have received amiodarone or other Vaughan Williams class I or III antiarrhythmic drugs in the last 6 months, untreated/poorly controlled hypothyroidism, hyperthyroidism, acute or chronic hepatic failure, other requirements of antiarrhythmic drug therapy, recent cardiac surgery in the preceding 30 days, and those who are pregnant.

Intervention: Patients aged 18 years or older who develop new-onset atrial fibrillation in the setting of severe sepsis or septic shock and in whom the medical team deems appropriate to initiate amiodarone therapy in will be considered for study inclusion. All patients will receive a 150 mg IV bolus dose of amiodarone, followed immediately by a continuous infusion of 1 mg/min for the first six hours, with a recommended reduction to 0.5 mg/min subsequently. Conversion from IV to PO amiodarone will occur based on patient hemodynamic stability and physician/pharmacist discretion. Patients will be randomized to receive amiodarone at a full loading dose (≥ 5g IV or ≥10g PO +/- 20%) or a partial loading dose (<4g IV or < 8g PO). The assigned total loading dose will include all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO amount (accounting for 50% bioavailability of PO versus IV amiodarone). The primary attending or fellow physician may over-ride randomization if the patient's amiodarone dose if the patient's severity of illness warrants a duration that differs from that assigned during randomization. In the full loading dose group, discontinuation of amiodarone will be at the discretion of the physician/pharmacists, after the pre-determined randomization loading dose has been provided.

Management Components: Facilities to be used throughout the project include the University Hospital and The University of Texas Health Science Center at San Antonio. Equipment use for direct patient care will be in keeping with standards-of-care, without any additional equipment being required for the clinical research study.

Data Collection: Data collection will include age, race, gender, body mass index (BMI), data for calculating an Acute Physiology and Chronic Health Evaluation (APACHE II) and Sequential Organ Failure Assessment (SOFA) scores, suspected source of infection, identified pathogens, pre-existing conditions that may predispose the patient to AF and the severity/classification of such illness (coronary artery disease, heart failure, chronic kidney disease, chronic obstructive pulmonary disease, diabetes mellitus); vital signs at the onset of AF (mean arterial pressure, systolic blood pressure, heart rate), lactate, pH (scale of acidity), and serum bicarbonate at the time of AF onset; fluid resuscitation volume for the 24 hours prior to AF, vasopressor use (including drug, dose, duration) in the preceding 24 hours; other medications used to stabilize hemodynamic status in AF (e.g. β-blockers, calcium channel blockers, digoxin), other attempted methods of cardioversion attempted prior to amiodarone use (e.g. direct current cardioversion, other antiarrhythmic drug therapy); amiodarone loading dose, cumulative study amiodarone dose; the duration of time spent in AF before conversion to normal sinus rhythm (NSR), the incidence of AF recurrence; and hemodynamic variables to be assessed at various time points after the initiation of amiodarone (-6 hours, at onset of AF, 2 hours, 6 hours, 12 hours, and every 6 hours thereafter until day 7 or death) including mean arterial pressure, central venous pressure, systolic blood pressure, heart rate, pH, serum bicarbonate, and serum lactate.

Monitoring for Efficacy and Safety:

Efficacy: Patients will be stratified based on response to therapy into one of three groups: conversion to NSR, non-converting AF that is hemodynamically stable or non-converting AF that is hemodynamically unstable. The primary efficacy outcome is the mean heart rate every 6 hours after initiation of the amiodarone infusion to day 7 or death. Secondary efficacy endpoints will include the percentage of time spent hemodynamically unstable in the first 7 days following amiodarone initiation, ICU LOS, hospital LOS and 28-day mortality along with comparisons of the individual portions of the hemodynamic endpoints [mean arterial pressure (MAP), heart rate (HR), systolic blood pressure(SBP)], cumulative vasopressor doses of norepinephrine and vasopressin, central venous pressure (CPR), conversion to NSR, maintenance of NSR, proportion of time spent in NSR after the start of the infusion to day 7 or death, pH, standard bicarbonate, serum lactate, and central venous oxygen saturation.

Safety: Safety outcomes include worsening of hypotension (largely related to the rate of infusion and the polysorbate 80 diluent), bradycardia, acute elevations of liver function tests ≥ 3 times the upper limit of normal, phlebitis, QTc prolongation, skin reactions, neuropathy, and pulmonary toxicity. We will also collect premature study discontinuation due to any adverse event. Because the experimental group of this study is a partial load of amiodarone, rather than a full load, it is likely that the experimental group will experience fewer amiodarone related adverse effects than those receiving the current practice. In the setting of worsening hemodynamic stability during amiodarone infusion (i.e. SBP <90 mmHg OR MAP < 70 mmHg, despite HR control of < 120 bpm; need for fluid boluses ± vasopressors or dobutamine), which the medical team believes to be caused by IV amiodarone therapy:

1. the amiodarone infusion rate should be decreased by 50%, with efforts to increase back to the standard infusion rate after the patient is hemodynamically stable, or
2. switch from IV amiodarone to PO amiodarone therapy at a dose of 400 mg PO three times daily (TID), or
3. emergent electro-cardioversion at the discretion of the medical team (as is the standard of care)

Data Analysis Plan: Data will be collected and stored using Microsoft Excel or Access. After data organization and cleaning, data will be imported into JMP 12.0 or SPSS. Data will be analyzed using both descriptive and comparative statistics. The primary outcome will be analyzed using repeated measures ANOVA. Nominal and ordinal variables will be compared using Chi-square test or Fisher's Exact test, as appropriate. Continuous variables will be tested for normality using the Shapiro-Wilk W goodness of fit test. Continuous variables with normal distributions will be compared using the student's t-test, while non-parametric variables will be compared using the Wilcoxon rank sum test. Statistical significance will be defined as an alpha level less than 0.05.

All baseline demographics, including patient comorbidities, amount of fluid resuscitation, previous vasoactive therapies, and use of other interventions such as direct current cardioversion, will be entered into a multivariate regression model if the p value is less than 0.20 on univariate comparison between treatment groups. The multivariate regression model will be used to assess if baseline factors or previous treatment other than the intervention affected the study outcomes.

Based on extrapolation from available literature assessing HR control at 24 hours, we estimate that the full loading dose group will have a mean HR of 110 bpm over the course of 7 days, while the partial loading dose group will have a mean HR of 130 bpm over the course of 7 days. 7 day mean HR that is 20 bpm lower than the partial loading dose group. Therefore, we estimate that 250 patients will be necessary in each group to have an 85% power to detect a difference, assuming a 15% drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* New onset atrial fibrillation
* Severe sepsis or septic shock (defined by ≥2 systemic inflammatory response syndrome criteria + infection)

Exclusion Criteria:

* Age < 18 years
* History of atrial flutter
* History of atrial fibrillation
* QTc >500 msec at baseline
* 2nd or 3rd degree AV block
* Currently receiving anti-arrhythmic therapy
* Untreated thyroid dysfunction
* Acute or chronic hepatic failure
* Other indication for antiarrhythmic therapy
* Recent cardiac surgery in last 30 days
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05; Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany A Kalich, Principal Investigator — UT Health San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Partial Load: 150 mg intravenous (IV) bolus dose of amiodarone, followed immediately by continuous infusion 1 mg/min for 6 hours, with a reduction to 0.5 mg/min subsequently. Conversion from IV to oral (PO) amiodarone will occur based on patient hemodynamic stability and physician/pharmacist discretion. Patients will receive <4g IV or < 8g PO. The assigned total loading dose will include all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO amount (accounting for 50% bioavailability of PO versus IV amiodarone).
  Amiodarone: Patients will receive a 150 mg IV bolus amiodarone dose, followed by a 1 mg/min continuous infusion for six hours, then 0.5 mg/min. Conversion to PO amiodarone will be based on patient hemodynamic stability and physician/pharmacist discretion. The total loading dose will be calculated based on all IV and PO amiodarone
- Full Load: All patients will receive a 150 mg intravenous (IV) bolus dose of amiodarone, followed immediately by a continuous infusion of 1 mg/min for the first six hours, with a recommended reduction to 0.5 mg/min subsequently. Conversion from IV to oral (PO) amiodarone will occur based on patient hemodynamic stability and physician/pharmacist discretion. Patients randomized to the partial load arm will receive (≥ 5g IV or ≥10g PO +/- 20%). The assigned total loading dose will include all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO amount (accounting for 50% bioavailability of PO versus IV amiodarone).
  Amiodarone: Patients will receive a 150 mg IV bolus amiodarone dose, followed by a 1 mg/min continuous infusion for six hours, then 0.5 mg/min. Conversion to PO amiodarone will be based on patient hemodynamic stability and physician/pharmacist discretion. The total loading dose will be calculated based on all IV and PO
Period: Overall Study
Arm/Group | Partial Load | Full Load
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Partial Load: 150 mg intravenous (IV) bolus dose of amiodarone, followed by continuous infusion of 1 mg/min for 6 hours, with recommended reduction to 0.5 mg/min. Conversion from IV to oral (PO) amiodarone will occur based on patient hemodynamic stability and physician/pharmacist discretion. Patients randomized to the partial load arm will receive <4g IV or < 8g PO. The assigned total loading dose will include all IV and PO amiodarone administered within 7 days from initiation of amiodarone. All doses will be compared in total PO amount (accounting for 50% bioavailability of PO versus IV amiodarone).
  Amiodarone: Patients will receive a 150 mg IV bolus amiodarone dose, followed by a 1 mg/min continuous infusion for six hours, then 0.5 mg/min. Conversion to PO amiodarone will be based on patient hemodynamic stability and physician/pharmacist discretion. The total loading dose will be calculated based on all IV and PO amiodarone
- Total: Total of all reporting groups
Arm/Group | Partial Load | Full Load | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.21 (16.5) | 54.8 (10.27) | 62 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean HR Every 6 Hours Within the First 7 Days
Description: Evaluate two amiodarone dosing strategies, a full loading dose versus a partial loading dose, in patients with new-onset atrial fibrillation (AF) due to severe sepsis or septic shock to assess the effect on:
  • Mean heart rate every 6 hours within the first 7 days following initiation of amiodarone
Time Frame: 7 days
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Groups:
- Partial Load: < 10g oral loading dose of amiodarone
- Full Load: 10 g (+/- 20%) oral loading dose of amiodarone
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
Beats per minute
  Average heart rate measured every 6 hours | 115 (16) | 122 (20)
  Average heart rate measured at 7 days | 71 (8) | 94.5 (9.5)

2. Secondary Outcome: Percentage of Time Spent Hemodynamically Unstable After Initiation of Amiodarone Infusion to Day 7 or Death
Description: Hemodynamic instability: 1. SBP <90 mmHg OR MAP < 70 mmHg AND HR ≥ 120 bp for ≥ 2 hours OR 2. HR ≥ 120 for ≥ 2 hours OR 3. Fluid boluses ± vasopressors or dobutamine. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 39 | 11

3. Secondary Outcome: Percentage of Time of Conversion to Normal Sinus Rhythm
Description: Percentage of time patients spent with conversion from atrial fibrillation to normal sinus rhythm. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 100 | 100

4. Secondary Outcome: Percentage of Time Patients Spent in Atrial Fibrillation
Description: Percentage of time in atrial fibrillation vs normal sinus rhythm or other during a 7 day period. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 82 | 65

5. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: Mean arterial pressure (MAP) measured over 7 days
Time Frame: 7 days
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
mmHg | 64 [60 to 73] | 75 [17 to 89]

6. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: Systolic blood pressure (SBP) measured over 7 days
Time Frame: 7 days
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
mmHg | 108 [89 to 114] | 124 [99 to 135]

7. Secondary Outcome: Heart Rate (HR)
Description: Heart rate (HR) measured over 7 days
Time Frame: 7 days
Measure: Mean (Full Range); unit: Beats per minute
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
Beats per minute | 70 [66 to 80] | 85 [78 to 110]

8. Secondary Outcome: Percentage Time of Vasopressor Norepinephrine Use
Description: Percentage time of Use of the vasopressor Norepinephrine in addition to the amiodarone. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 5
percentage of time | 80 | 75

9. Secondary Outcome: Percentage Time of Vasopressor Vasopressin Use
Description: Percentage time of use of the vasopressor Vasopressin in addition to amiodarone. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 40 | 25

10. Secondary Outcome: Percentage of Time of Vasopressor Phenylephrine Use
Description: Percentage of time of use of the vasopressor Phenylephrine in addition to amiodarone. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 0 | 50

11. Secondary Outcome: Percentage of Time of Corticosteroid Use
Description: Percentage of time of use of a corticosteroid for treatment in addition to amiodarone use. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 20 | 25

12. Secondary Outcome: Percentage of Time of Dobutamine Use
Description: Percentage of time of use of Dobutamine in addition to amiodarone intervention. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 0 | 0

13. Secondary Outcome: Percentage of Time of Concomitant Rate Control Medication Use
Description: Percentage of time of Additional medications used to control heart rate in addition to amiodarone. The reported data represents a cumulative percentage of time for the entire group of participants.
Time Frame: 7 days
Measure: Number; unit: percentage of time
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
percentage of time | 20 | 75

14. Secondary Outcome: Concomitant Rhythm Control Medication or Intervention Use
Description: Use of additional medications used with amiodarone to control heart rhythm.
Time Frame: 7 days
Population: Outcome measure data were not collected or analyzed for this outcome, study terminated early due to lack of funding and due to Investigator leaving institution
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: 28-day Mortality
Description: Survival to 28 days post initiation of treatment.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
participants | 4 | 1

16. Secondary Outcome: Intensive Care Unit Length of Stay (ICU LOS)
Description: Number of days spent in intensive care unit after admission.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Partial Load | Full Load
Number analyzed (Participants) | 5 | 4
days | 6.5 [3.5 to 14.75] | 6 [5 to 28]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Partial Load | Full Load
All-Cause Mortality (participants affected / at risk) | 4/5 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT02668432/Prot_SAP_000.pdf